CLINICAL TRIAL: NCT00036075
Title: Study Using CP-461 to Treat Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Cell Pathways (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI-461-006
Record Dates: First submitted 2002-05-07; First posted 2002-05-08 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — (5-fluoro-2-methyl-1-(4-pyridyl)methylene-3-(N-benzyl)-indene)-acetamide hydrochloride

INTERVENTIONS:
Drug: CP-461

SUMMARY:
The purpose of this study is to investigate whether an investigational drug, CP-461, is safe and effective for the treatment of patients with prostate cancer and who have measurable disease.

ELIGIBILITY:
Eligibility Criteria:

* Male 18 years of age.
* Histologically confirmed adenocarcinoma of the prostate, stage D1 or D2.
* Failure of androgen ablation (orchiectomy or LHRH, flutamide).
* Patients must have PSA progression and progression in measurable disease.
* No prior history of systemic chemotherapy.
* No investigational drugs within 4 weeks of study entry.
* No radiation therapy or hormonal therapy within 4 weeks of study entry.
* No isotope therapy within 6 weeks of study entry.
* No antiandrogens within 4 weeks of study entry. Patients must continue LHRH.
* If patients had prior surgery, it must be at least 21 days prior to study entry, and the patient must have recovered from all side effects.
* Patients must have stopped bisphosphonates 28 days prior to study entry.
* No prior malignancy allowed except for adequately treated basal cell or squamous cell skin cancer, or adequately treated stage I or II cancer from which the patient is currently in remission, and has been disease free for at least 5 years.
* Patients must have recovered from major infections and/or surgical procedures, and in the opinion of the investigator not have significant active concurrent medical illness, such as a history of significant neurologic or psychiatric disorders including psychotic disorders, dementia, or seizures that would preclude protocol treatment or survival.
* All patients must be informed of the investigational nature of the study and must sign and give written informed consent in accordance with institutional and federal guidelines.
* No other chemotherapeutic, biological response modifiers, radiation therapy, corticosteroid therapy, or hormonal concomitant therapy (except continuation of LHRH) may be given during treatment. Patients should not be planning on receiving concomitant bisphosphonates.
* ECOG Performance Status = 0-3.
* WBC > or = 3500/ul or ANC > or = 1500/ul.
* Bilirubin < or = ULN.
* Creatinine < or = 2.0 mg/dl.
* Platelets > or = 100,000/ul.
* ALT or AST < 2.5 X ULN.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2001-08; Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Columbia Presbyterian Medical Center, New York, New York
  - University of Washington, Seattle, Washington